CLINICAL TRIAL: NCT06550492
Title: In Reducing the Negative Effects of Surgical Conditions Comparison of Two Different Methods: Use of Double Layer Mask Against Smoke Filtering Electrocautery
Brief Title: Reducing the Negative Effects of Surgical Conditions Use of Double Layer Mask Against Electrocautery With Smoke Filter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Nurhan Bagacli, Chief Researcher, Ataturk University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: AtaturkU25
Record Dates: First submitted 2024-08-05; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Surgical Procedure, Unspecified
Keywords: surgical smoke
MeSH Terms: interventions — Double-Blind Method

STUDY DESIGN:
Intervention Model Description: experimental group using smoke filtering electrocautery device, experimental group using double mask and control group using single mask
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- experimental group using smoke filtering electrocautery device (Experimental): experimental group using smoke filtering electrocautery device
  Interventions: Device: smoke filtering electrocautery device
- experimental group using double mask (Experimental): experimental group using double mask
  Interventions: Other: double mask
- control group (No Intervention): group using standard methods

INTERVENTIONS:
Device: smoke filtering electrocautery device — A smoke-filtering electrocautery device was used during surgery.
  Arms: experimental group using smoke filtering electrocautery device
Other: double mask — A double-layer mask was used during the operation.
  Arms: experimental group using double mask

SUMMARY:
This study was conducted to determine and compare the effectiveness of the smoke filtering electrocautery device used to reduce the negative effects of surgical smoke and the use of a double layer mask.

DETAILED DESCRIPTION:
The research was conducted as a randomised controlled experimental study. The research was collected between November 2023 and February 2024 in Atatürk University Health Research and Application Centre Operating Theatre unit. Data were collected using the Personal Information Form, Specified Health Problems Questionnaire, and the Practice Record Form to record blood gas laboratory results. The study was conducted with 90 (30 control, 30 double mask, 30 device) operating theatre workers. The population of the study consisted of Atatürk University Health Practice and Research Hospital Operating Theatre unit employees between November 2023 and February 2024. In this study, a priori power analysis was performed to determine the sample size. In the power analysis, the sample of the study consisted of a total of 90 people, 30 people in the group using cautery device with smoke filtering system, 30 people in the group using double masks and 30 people in the control group, with an effect size of 0.5%, which is the medium effect size according to Cohen, an error margin level of 0.05% and a confidence interval of 0.95%, with a 95% population representativeness.

ELIGIBILITY:
Inclusion Criteria:

* people over the age of 18.
* People who agreed to participate in the study,
* who have been working in the operating theatre for at least one year.
* people who do not have chronic diseases Voluntary personnel who volunteered to co-operate were included in the study.

Exclusion Criteria:

* People who did not agree to participate in the study,
* persons who have been working in the operating theatre for less than one year
* people with chronic diseases,
* people who withdrew from the study before all data were collected
* Personnel whose laboratory results could not be analysed were excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Application Registration Form | 1 day
  This form includes laboratory findings such as COHb, MetHb, PaO2, PaCO2, pH, HCO3, SpO2, Hg that may be affected in the person exposed to surgical smoke. In the study, it was examined whether exposure to surgical smoke affected these values.
Questionnaire on Reported Health Problems | 1-2 day
  The questionnaire form, which was created by the researcher by reviewing the literature on the subject, includes 45 health problems that may occur in the short term as a result of exposure to surgical smoke and a scale related to the frequency of experiencing these problems. in the questionnaire, the every day option shows the maximum value, the never option shows the minimum value

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Karaman Özlü, Professor, Study Director — zkaraman@atauni.edu.tr
Locations (1):
- Atatürk University Health Application and Research Centre, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Karaman Özlü Z., Uymaz Aras G., Bayrak A. (2022). Ameliyathanedeki Görünmez Tehlike: Cerrahi Duman. Arşiv Kaynak Tarama Dergisi, 31(1),10-14. doi:10.17827/aktd.969260 — https://dergipark.org.tr/en/pub/aktd/article/969260